CLINICAL TRIAL: NCT02368249
Title: Does Terlipressin Improve Renal Outcome After Liver Surgery - A Double-Blinded Randomized Control Trial (TIROL-Trial)
Brief Title: Does Terlipressin Improve Renal Outcome After Liver Surgery
Acronym: TIROL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no focus on this topic
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ksenija Slankamenac, MD PhD, University of Zurich
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2012-0581
Record Dates: First submitted 2015-02-09; First posted 2015-02-23 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Terlipressin; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients receiving post-operative placebo (Ringer lactate solution) treatment to preserve the renal function
  Interventions: Drug: Placebo
- Terlipressin Group (Experimental): Patients receiving a post-operative intravenous terlipressin treatment in association with human albumin to preserve the renal function
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — Patients are receiving a post-operative intravenous terlipressin treatment in association with human albumin to preserve the renal function
  Other Names: Gylpressin
  Arms: Terlipressin Group
Drug: Placebo — Patients are receiving a post-operative intravenous Ringer's lactate solution
  Other Names: Ringer's lactate solution
  Arms: Control Group

SUMMARY:
The investigators aim to address whether terlipressin improves the renal outcome after liver surgery. Therefore the investigators are planning to conduct a double-blinded randomized control trial. The investigators will randomize patients undergoing any kind of liver surgery and being at increased moderate to high risk for post-operative acute renal failure into a control group receiving post- operative a placebo or into a group receiving post-operatively terlipressin in combination with human albumin.

ELIGIBILITY:
Inclusion Criteria:

* >=12% risk for post-operative ARF on our recently developed and validated prediction score for ARF after liver surgery, patients will need five points or more in the pre-operative assessment of the predictors to be enrolled in the trial

Exclusion Criteria:

* < 18 years
* liver cirrhosis
* coronary insufficiency with ST-elevation or ST-depression in the - - intra-operative ECG as signs of an acute coronary syndrome
* pregnancy and breast feed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
serum creatinine peak level within 48 hours post-operative | within 48 hours post-operative

SECONDARY OUTCOMES:
the urinary output/24h | Post Operative Day 0 to 3
Need for hemofiltration and/or hemodialysis | Post Operative Day 0 - 14
  participants will be followed for the duration of hospital stay, an expected average of 14 days
Morbidity & mortality | Post Operative Day 0 - 14
  measured by the comprehensive complication index; participants will be followed for the duration of hospital stay, an expected average of 14 days
Liver function | Post Operative Day 0 - 5
  assessed by serum levels of aspartate aminotransferase (AST) and alanine aminotransferase (ALT)
length of hospital stay | Post Operative Day 0 - 14
  in days; participants will be followed for the duration of hospital stay, an expected average of 14 days
length of ICU stay | Post Operative Day 0 - 7
  in days; participants will be followed for the duration of ICU stay, an expected average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alain Clavien, MD PhD, Study Director — Departement of Visceral and Transplantation Surgery Zurich
Locations (1):
- Department of Visceral and Transplantation Surgery of the University Hospital of Zurich, Zurich, Switzerland